CLINICAL TRIAL: NCT05135949
Title: Strength and Function After Non-operative Treatment of Displaced Olecranon Fractures in the Elderly: Implications of Standing UP From a Seat
Brief Title: Strength After Elbow Fractures in the Elderly
Acronym: STAND-UP
Status: Recruiting | Type: Observational
Sponsor: Fraser Orthopaedic Research Society (Network)
Responsible Party: Sponsor
Other Study IDs: 2020-147
Record Dates: First submitted 2021-11-04; First posted 2021-11-26 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Fracture;Elbow
Keywords: Operative; Non Operative
MeSH Terms: conditions — Elbow Fractures | interventions — Patient Reported Outcome Measures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Operative: Internal fixation of the displaced olecranon fracture.
  Interventions: Other: Patient Reported Outcomes; Other: Strength Test
- Non Operative: Conservative treatment as determined by the treating surgeon.
  Interventions: Other: Patient Reported Outcomes; Other: Strength Test

INTERVENTIONS:
Other: Patient Reported Outcomes — Satisfaction, Disabilities of the Shoulder, Arm and Hand
Other: Strength Test — Handheld dynamometer to measure tricep extension

SUMMARY:
Elderly patients strength and function, specifically the ability to rise from a seat after either operative or non operative treatment of an mayo type 2 olecranon fracture.

DETAILED DESCRIPTION:
Elderly patients with an olecranon fracture will receive appropriate treatment as determined by the treating surgeon. Patients will then be assessed at 6 weeks, 6 months and 12 months post treatment. Assessments include, range of motion, patient reported outcomes and a strength test.

ELIGIBILITY:
Inclusion Criteria:

1. ≥65 years of age
2. Mayo type II olecranon fracture
3. Ambulatory (with or without the use of walking aides)

Exclusion Criteria:

1. Additional injuries to the affected arm or contralateral arm
2. Associated nerve injury
3. Dementia or cognitive impairment that inhibits the collection of outcome measures
4. Likely problems, in the judgement of the investigator, with maintaining follow-up (i.e. patients with no fixed address, not mentally competent to give consent, intellectually challenged, patients without adequate support, etc.)
5. Injury or previous deficit to the contralateral arm
6. Currently enrolled in any other research study involving drugs or medical devices
7. Open fractures
8. Inability to provide informed consent

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: Elderly patients for displaced olecranon fractures
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-02-22 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Extension Strength | 12 Months
  Patients will push down on their distal forearm through a hand held dynamometer, to measure tricep extension strength

SECONDARY OUTCOMES:
Arc of Motion | 12 months
  Elbow extension and elbow flexion measured with a goniometer
Mayo Elbow Performance Index | 12 Months
  An instrument used to test the limitations, caused by pathology, of the elbow during activities of daily living. Higher scores indicate a better outcome.
Disabilities of the Arm, Shoulder, and Hand | 12 Months
  A 30 Item questionnaire that measures an individuals' ability to complete tasks, absorb forces and severity of symptoms. Lower scores will indicated better outcomes.Lower scores will indicate better outcomes.
Satisfaction Score | 6 weeks, 6 months and 12 months
  Soccer out of 10, higher the score the better the outcome

CONTACTS AND LOCATIONS:
Overall Officials: Farhad Moola, PhD, Principal Investigator — Orthopaedic Surgeon
Locations (1):
- Royal Columbian Hospital, New Westminster, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-08): https://cdn.clinicaltrials.gov/large-docs/49/NCT05135949/Prot_SAP_000.pdf